CLINICAL TRIAL: NCT05377944
Title: A Multicenter, Randomized, Double-Blind, Parallel-Arm, Phase 3 Study to Compare Efficacy and Safety of BAT2306 With Cosentyx® in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Assessment on Efficacy and Safety of BAT2306 and Cosentyx® in Plaque Psoriasis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAT-2306-002-CR
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-10

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT2306 (Experimental): Patients will receive subcutaneous treatment of 300 mg BAT2306 (2 injections of 150 mg/1 ml) via PFS at weeks 0, 1, 2, 3, and 4 followed by dosing every 4 weeks, thereafter up to Week 40.
  Interventions: Drug: BAT2306
- EU-approved Cosentyx (Active Comparator): Patients will receive subcutaneous treatment of 300 mg EU-approved Cosentyx (2 injections of 150 mg/1 ml) at weeks 0, 1, 2, 3, and 4 followed by dosing every 4 weeks, thereafter up to Week 40.
  Interventions: Drug: EU-approved Cosentyx

INTERVENTIONS:
Drug: BAT2306 — 150 mg/1 ml/injection (2 injections/visit)
  Other Names: Recombinant human monoclonal antibody against IL-17A
  Arms: BAT2306
Drug: EU-approved Cosentyx — 150 mg/1 ml/injection (2 injections/visit)
  Other Names: secukinumab injection
  Arms: EU-approved Cosentyx

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel-arm, Phase 3 study designed to compare efficacy, safety, immunogenicity, and PK of BAT2306 with Cosentyx in patients with moderate to severe plaque psoriasis.

The study is composed of a ≤ 28-day screening period, a 24-week initial treatment period (Treatment Period 1 [TP1]), and a 28-week secondary treatment period (Treatment Period 2 [TP2]). The study will be a maximum of 56 weeks.

DETAILED DESCRIPTION:
Primary objective:

• To demonstrate equivalent efficacy of BAT2306 and Cosentyx® in patients with moderate to severe plaque psoriasis.

Secondary objectives:

* To evaluate the efficacy of BAT2306 compared with Cosentyx over the study period based on secondary efficacy endpoints.
* To evaluate the safety and tolerability of BAT2306 compared with Cosentyx over the study period.
* To evaluate the immunogenicity of BAT2306 compared with Cosentyx over the study period.
* To evaluate the steady-state pharmacokinetics (PK) of BAT2306 compared with Cosentyx.
* To assess safety and immunogenicity after transition from Cosentyx to BAT2306.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old with a diagnosis of plaque-type psoriasis for at least 24 weeks before screening.
2. Have moderate to severe plaque-type psoriasis as defined at screening and baseline by:

   1. PASI ≥ 12,
   2. IGA ≥ 3 (based on a scale of 0-4), and
   3. BSA affected by chronic plaque-type psoriasis ≥ 10%
3. Candidates for systemic therapy, defined as having chronic plaque-type psoriasis considered inadequately controlled by:

   1. topical treatment and/or
   2. phototherapy and/or
   3. previous systemic therapy.
4. Female patients of childbearing potential and male patients with a female partner of childbearing potential must be willing to use a highly effective contraceptive precaution throughout the study period and continuing for at least 20 weeks after the last dose of study drug. See APPENDIX 1 for the acceptable highly effective contraceptive methods. Abstinence from heterosexual intercourse is accepted when this is the usual lifestyle of the patient and must be continued for at least 20 weeks after the last dose of study drug. A female patient is considered not of childbearing potential when postmenopausal (at least 12 consecutive months without menses without an alternative medical cause) or surgically sterilized (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy).
5. If female of childbearing potential, patient should have a negative pregnancy test result at screening and baseline visits.
6. Must be willing to provide written consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Have any forms of psoriasis at the time of the screening visit other than plaque-type such as erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis or other skin conditions (e.g., eczema) that would interfere with evaluations of the effect of investigational product on psoriasis.
2. Have previously received secukinumab, a biosimilar of secukinumab, or any drug that targets interleukin-17 or the IL-17 receptor (eg, ixekizumab, brodalumab).
3. Weight > 120 kg.
4. Have received any monoclonal antibody-based biologic drugs for the treatment of PsO or PsA or with a potential effect on the study condition, other than those prohibited (see exclusion #2) within 5 half-lives or 6 months, whichever is longer, before baseline visit.
5. Have received non-monoclonal antibody biological drugs (eg, etanercept) for the treatment of PsO or PsA within 12 weeks or 5 half-lives (whichever is longer) before baseline visit.
6. Have received topical therapies for the treatment of psoriasis (such as corticosteroids, vitamin D analogs, retinoids, herbal or non-pharmacological topical preparations other than moisturizers or emollients) within 2 weeks before baseline visit.

And so on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | 0-8 weeks(EMA, PMDA) or 0-12 weeks(FDA, NMPA)
  * EMA, PMDA, and Agencies other than the FDA and NMPA: Percent change from baseline in Psoriasis Area and Severity Index (PASI) score to Week 8
  * FDA and NMPA: Percent change from baseline in PASI score to Week 12
  Minimum value 0, maximum value 72. Higher score means worse outcome.

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) score | Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Percentage change from baseline in PASI score at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44. Minimum value 0, maximum value 72. Higher score means worse outcome.
PASI-50/75/90/100 | Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Proportion of patients who achieve at least 50/75/90/100% improvement from baseline in PASI (PASI-50/75/90/100) at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44.
  Higher score means better outcome
Investigator's Global Assessment (IGA) | Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44
  Change from baseline in Investigator's Global Assessment (IGA mod 2011) at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, and 44. Minimum value 0, maximum value 4. Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No